CLINICAL TRIAL: NCT02664753
Title: L-carnitine as an Adjunct Treatment for Septic Shock Patients With Acute Kidney Injury: a Multicentre, Randomized, 2-parallel Group, Superiority Trial
Brief Title: L-carnitine as an Adjunct Treatment for Septic Shock Patients With Acute Kidney Injury
Acronym: CarniSave
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Exposure to serious adverse events related to the research (i.e., death), the mnts = 54% versus 58 deaths out of 121 patients = 48%).onitoring committee unanimously recommended discontinuation of the trial.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-N/2015/PR-01
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Severe Sepsis; Shock, Septic; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Carnitine group (Experimental): Patients in the experimental arm will receive 10 days of intravenous L-carnitine treatment followed by 46 days of oral L-Carnitine treatment.
  Intervention: 56 days of weight-adjusted L-Carnitine treatment
  Interventions: Drug: 56 days of weight-adjusted L-Carnitine treatment
- Placebo then open group (Placebo Comparator): Patients in the placebo arm will receive 10 days of intravenous isotonic saline in a fashion analogous to the experimental arm (they study is thus blinded for the first 10 days and then open there afterwards).
  Intervention: 10 days of intravenous placebo (isotonic saline)
  Interventions: Drug: 10 days of intravenous placebo (isotonic saline)

INTERVENTIONS:
Drug: 56 days of weight-adjusted L-Carnitine treatment — Patients in the experimental arm will receive 10 days of intravenous L-carnitine treatment followed by 46 days of oral L-Carnitine treatment.
  Day 1: a first bolus of 6g of L-Carnitine is administered with a syringe driver of 50 ml.
  Day 2 to Day 10: Two mini-perfusions are prepared each day, corresponding to 1 administration every 12 hours. 50 mg/kg/day (rounded up to the next gram) L-Carnitine is added to each syringes
  For the next 46 days, patients will take oral doses of L-Carnitine as follows:
  < à 60kg : 2g/day > 60kg : 3g/day If the patient leaves the hospital before D10, oral treatment can be initiated at the end of the hospitalization
  Arms: L-Carnitine group
Drug: 10 days of intravenous placebo (isotonic saline) — Patients in the placebo arm will receive 10 days of intravenous isotonic saline in a fashion analogous to the experimental arm (they study is thus blinded for the first 10 days and then open there afterwards).
  Day 1: 1 50ml syringe driver of 50 ml isotonic saline solution . Day 2 to Day 10 : Two syringe drivers of 50 ml of isotonic saline solution are prepared each day, one during the morning and one during the evening.
  Arms: Placebo then open group

SUMMARY:
The primary objective of this study is to compare 28 day mortality rates between septic shock patients with acute renal insufficiency treated via L-Carnitine (as an adjunct therapy) versus a similar group of patients not receiving L-Carnitine adjunct therapy.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. First secondary objective of this study is to compare 10 day mortality rates of septic shock patients with renal insufficiency treated via L-Carnitine (as an adjunct therapy) for 56 days versus a patients not receiving L-Carnitine adjunct therapy

B. To compare study arms in terms of patient safety.

C. To compare study arms in terms of further clinical outcomes, with special emphasis on nephrological outcomes.

D. To study (and compare between arms) the kinetic curves of free and total serum carnitine. Renal replacement therapy rapidly depletes the body's carnitine levels. Tracking adequate carnitine levels is therefore important for the interpretation of study results.

E. To constitute a bio-bank in association with the study for future ancillary studies (e.g. kidney injury marker studies, carnitine-responders versus non-responders, and other exploratory studies.

ELIGIBILITY:
Inclusion Criteria:

* • The emergency inclusion procedure was correctly applied according to French law (signature of consent form by a patient-designated trusted person or a family member, or a medical decision to proceed with patient inclusion if the latter two persons are unavailable) ---- OR ---- signature of the consent form by the patient

  * The patient must be insured or beneficiary of a health insurance plan
  * The patient is at least 18 years old
  * The patient was admitted to an intensive care unit (participating in the study) for sepsis or septic shock and presented with acute renal failure requiring, at some point, the use of extra-renal purification.
  * • The patient has sepsis or septic shock according to international criteria SEPSIS 3 (Singer et al, The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) ; JAMA. 2016)
  * The patient has acute renal insufficiency with an KDIGO score of 3
  * The patient has started continuous renal replacement therapy (CRRT) or intermittent renal replacement therapy (IRRT) within the previous 72 hours, or will start RRT (CRRT or IRRT) within the next 72 hours.

Exclusion Criteria:

* • The patient is participating in, or has participated in over the past three months, another interventional study that may interfere with the results or conclusions of this study

  * The patient is in an exclusion period determined by a previous study
  * The patient is under judicial protection, or is an adult under guardianship
  * The patient is pregnant, parturient or breastfeeding
  * The patient is susceptible to procreate and does not use methods of effective contraception (contraceptive hormonal ring, surgical contraception, contraceptive implant, contraceptive pill, male or female sheaths, skin patch, intrauterine contraceptive device)
  * If the patient is unable to sign a consent form: the patient-designated trusted person or family member refuses to sign the consent form
  * If the patient is unable to sign a consent form: It is impossible to correctly inform the patient-designated trusted person or family member
  * The patient is able/apt to sign a consent form, but refuses to do so
  * The patient is able/apt to sign a consent form, but cannot be correctly informed
  * Septic shock without associated AKI
  * Patients with a known allergy to L-Carnitine or other component of levocarnil oral solution or for injection
  * Pre-existing chronic disease requiring dialysis
  * The patient has stage 4 CKD with baseline DFG (CDK) if known <30 ml
  * History of seizures or epilepsy
  * Chronic bowel disease or history of chronic diarrhoea
  * Under treatment with sodium valproate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days

SECONDARY OUTCOMES:
First secondary objective of this study is to compare 10 day mortality rates of septic shock patients with renal insufficiency treated via L-Carnitine (as an adjunct therapy) for 56 days versus a patients not receiving L-Carnitine adjunct therapy. | 10 days
  Mortality
Adverse Events per patient | 12 months (throughout study)
Survival | 12 months (throughout study)
The number of days alive and not on renal replacement therapy | 12 months
The number of days alive and free of renal failure | 12 months
The number of days alive and free of organ failure | 12 months
The number of days alive and not on mechanical ventilation | 12 months
The number of days alive and not in Intensive Care Unit (ICU) | 12 months
The number of days alive and not in hospital | 12 months
The number of days alive and free of (not requiring) catecholamines | 12 months
A vector of repeated measures of daily SOFA (Sequential Organ Failure Assessment score) scores available during the ICU stay | at ICU discharge (expected max of 28 days)
  Available daily scores will be aggregated into a vector for repeated measures analysis (similar to the agregation required for calculating a slope).
A vector of repeated measures of AKIN (Acute Kidney Injury Network score) score available during the ICU stay | at ICU discharge (expected max of 28 days)
  Available daily scores will be aggregated into a vector for repeated measures analysis (similar to the agregation required for calculating a slope).
A vector of repeated measures of serum creatinine | at ICU discharge (expected max of 28 days)
  Available measures will be aggregated into a vector for repeated measures analysis (similar to the agregation required for calculating a slope).
A vector of repeated measures of serum creatinine | at discharge from the nephrology department (expected max of 60 days)
  Available measures will be aggregated into a vector for repeated measures analysis (similar to the agregation required for calculating a slope).
A vector of repeated measures of lactate levels available during the ICU stay | at ICU discharge (expected max of 28 days)
  Available measures will be aggregated into a vector for repeated measures analysis (similar to the agregation required for calculating a slope).
Glomerular filtration rate (EpiCKD) | month 1
  (if the patient is on dialysis, the glomerular filtration rate is set at 0)
Glomerular filtration rate (EpiCKD) | month 2
  (if the patient is on dialysis, the glomerular filtration rate is set at 0)
Glomerular filtration rate (EpiCKD) | month 3
  (if the patient is on dialysis, the glomerular filtration rate is set at 0)
Glomerular filtration rate (EpiCKD) | month 6
  (if the patient is on dialysis, the glomerular filtration rate is set at 0)
Glomerular filtration rate (EpiCKD) | month 9
  (if the patient is on dialysis, the glomerular filtration rate is set at 0)
Glomerular filtration rate (EpiCKD) | month 12
  (if the patient is on dialysis, the glomerular filtration rate is set at 0)
Serum free carnitine level | baseline
Serum free carnitine level | after 48h of renal replacement therapy
Serum free carnitine level | day 7
Serum free carnitine level | day 14
Serum free carnitine level | month 1
Serum free carnitine level | month 2
Serum total carnitine level | baseline
Serum total carnitine level | after 48h of renal replacement therapy
Serum total carnitine level | day 7
Serum total carnitine level | day 14
Serum total carnitine level | month 1
Serum total carnitine level | month 2

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Reboul, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (11):
- France (11):
  - CHU de Caen, Caen
  - CH de Chartres, Chartres
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU Lyon, Lyon
  - CHU de Montpellier - Lapeyronie, Montpellier
  - CHU de Montpellier - St Eloi, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Poitiers, Poitiers
  - CHU de St Etienne, Saint-Priest-en-Jarez
  - CHU de Toulouse - Hôpital Rangueil, Toulouse

REFERENCES:
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500